CLINICAL TRIAL: NCT03522571
Title: Experimental Gingivitis in Patients With Altered Passive Eruption: A Case Control Study
Brief Title: Experimental Gingivitis in Patients With Altered Passive Eruption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rustam Aghazada (Other)
Responsible Party: Sponsor-Investigator, Rustam Aghazada, Principal Investigator, University of Roma La Sapienza
Organization: University of Roma La Sapienza (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: v. 01 02/12/2016
Record Dates: First submitted 2018-04-27; First posted 2018-05-11 (Actual); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Altered Passive Eruption of Teeth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with altered passive eruption - APE (Experimental): 3 teeth of the patients with altered passive eruption that will undergo to experimental gingivitis
  Interventions: Behavioral: Experimental gingivitis
- Patients with normal gingival anatomy - Non APE (Active Comparator): 3 teeth of the patients with normal gingival anatomy that will undergo to experimental gingivitis
  Interventions: Behavioral: Experimental gingivitis

INTERVENTIONS:
Behavioral: Experimental gingivitis — Individual cast models were prepared on alginate impressions. A 2-mm thick film of technical wax was set on the supra gingival area at buccal and proximal surfaces of study teeth on test quadrant. The stent were delivered at day 0. Subjects were instructed to wear the stent prior to the oral hygiene session throughout the experimental gingivitis period to prevent plaque removal during brushing of the remaining dentition. On Day 42 (T6): After recording of clinical parameters, oral hygiene instruction and an additional session of supragingival scaling, as needed, and polishing were given.

SUMMARY:
Altered passive eruption (APE) is an anatomical condition that is frequently diagnosed in periodontal clinical practice, especially for the ever-increasing demand of patients for the aesthetic improvement of their smile. In addition to its aesthetic value, however, altered passive eruption could also affect gingival and periodontal health. In fact, in the case of plaque accumulation, the altered passive eruption (APE) is likely to be a predisposing factor for a more rapid progression of gingivitis with higher inflammation indexes (Angulated Bleeding Score - AngBs and Modified Gingival Index - mGI). Notwithstanding, even if gingivitis in patients with altered passive eruption is developed much more rapidly, thorough home oral hygiene and plaque control conduces to complete clinical recovery. Further studies with a large number of patients are required to confirm the correlation between altered passive eruption and periodontal diseases.

DETAILED DESCRIPTION:
Study hypothesis

Despite the fact that many authors suggest that the patients with altered passive eruption are more susceptible to gingivitis and periodontitis due to the excess of gingiva, which impedes the correct oral hygiene procedure, there is to-date no clinical study confirming this assumption. The aim of the present study is therefore to examine the onset, progress and the healing of experimental gingivitis in patients with altered passive eruption when compared to patients with normal gingival anatomy.

Study design This is single centre interventional non randomised case-control study.

Interventions To achieve optimum gingival health and to standardize gingival baseline conditions all subjects participated in a pretrial period 7 days before T0. On day 7(T0), after professional scaling and polishing a powered toothbrush (Oral-B pro 3000, Braun, Procter and Gamble, USA), individually chosen interdental brush (Tepe, Sweden), and standard toothpaste (AZ - pro expert, Procter and Gamble, USA), along with oral hygiene instructions, were provided. Subjects were instructed to brush the teeth by using powered toothbrush.

Individual cast models were prepared on alginate impressions. A 2-mm thick film of technical wax was set on the supra gingival area at buccal and proximal surfaces of study teeth on test quadrant. The stent were delivered at day 0. Subjects were instructed to wear the stent prior to the oral hygiene session throughout the experimental gingivitis period to prevent plaque removal during brushing of the remaining dentition. On Day 42 (T6): After recording of clinical parameters, oral hygiene instruction and an additional session of supragingival scaling, as needed, and polishing were given.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* probing depth ≤ 3 mm

Exclusion Criteria:

* Smoking
* Periodontitis
* Systemic diseases
* Immunosuppressed or immunocompromised patients
* Use of medications affecting periodontal status
* Uncontrolled diabetes
* Pregnancy or lactation
* Addiction to alcohol or drugs
* Psychiatric problems
* Presence of any restorations on the examined quadrant
* Presence of periapical and endo-perio lesions
* Teeth with malposition and alteration in crown morphology
* Patients with an acute infection (abscess) in the site intended for treatment

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

PRIMARY OUTCOMES:
Change of Angulated bleeding score (AngBS) | Change of the value was assessed at T0, at day seven, fourteen, twenty-one, twenty-eight , thirty-five and at day forty-two
  Angulated bleeding score (AngBS) was introduced by Trombelli et al, which is a modification of the angulated bleeding index as reported by van der Weijden. After lightly drying the gingiva with compressed air, a periodontal probe (PCP 15 University of North Carolina(UNC), Hu Friedy, Chicago, Illinois, USA) was held at an angle of approximately 60° to the longitudinal axis of the tooth and in contact with the sulcular gingival tissues.
  Angulated bleeding score (AngBS) was scored as:
  0: no bleeding;
  1. bleeding upon probe stimulation;
  2. spontaneous bleeding.
Change of Gingival index (MGI) | Change of the value was assessed at T0, at day seven, fourteen, twenty-one, twenty-eight , thirty-five and at day forty-two
  Gingival index (MGI) according to Silness & Loe, but without probing component, due to not disturb plaque accumulation, was registered as:
  1. - Normal gingiva;
  2. - Mild inflammation - slight change in color and slight edema
  3. - Moderate inflammation - redness, edema and glazing,
  4. - Severe inflammation - marked redness and edema, ulceration with tendency to spontaneous bleeding.

SECONDARY OUTCOMES:
Plaque index (PLI) | Value was assessed at T0, at day seven, fourteen, twenty-one, twenty-eight , thirty-five and at day forty-two
  Plaque index (PLI), according to Silness & Loe was scored as:
  1. - No plaque ;
  2. - A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution
  3. - Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  4. - Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Quigley Hein Plaque Index (QH) | Value was assessed at T0, at day seven, fourteen, twenty-one, twenty-eight , thirty-five and at day forty-two
  Quigley Hein Plaque Index - QH (Modified by Turesky et al.) was registered after using disclosing solution as:
  0 - No plaque
  1. - Separate flecks of plaque at the cervical margin of the tooth
  2. - A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth
  3. - A band of plaque wider than one mm but covering less than one-third of the crown of the tooth
  4. - Plaque covering at least one-third but less than two-thirds of the crown of the tooth
  5. - Plaque covering two-thirds or more of the crown of the tooth
Gingival crevicular fluid volume (GCF) | Value was assessed at T0, at day seven, fourteen, twenty-one, twenty-eight , thirty-five and at day forty-two
  Gingival crevicular fluid volume (GCF), collected as previously described and measured according to Periotron 8.000 manufacturer's (OraFlow Inc., Plainview, New York, USA) instructions. The individual site was gently air dried in an apico-coronal direction without removal of any visible supragingival plaque. The area was carefully isolated with cotton rolls, to avoid salivary contamination. A sterile paper strip (Periopaper; OraFlow Inc.) was introduced into the crevice until mild resistance was felt. Attention was paid to avoid any mechanical injury to marginal tissues. The strip was left in place for 5 s and immediately transferred, for volume determination, to the calibrated, chair-side located Periotron 8,000 (OraFlow Inc.). Paper strips contaminated by gingival bleeding during gingival crevicular fluid (GCF) determination were discarded and corresponding data were recorded as missing.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, MD, DDS, MSc, Study Chair — University of Roma La Sapienza
Locations (1):
- Dipartimento di Scienze Odontostomatologiche e Maxillo Facciali, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF